CLINICAL TRIAL: NCT00485810
Title: A Study Examining Clinical Therapeutic Dose of Rapid Acting Intra-Muscular Olanzapine in Japanese Agitated Patients With Schizophrenia
Brief Title: Examining Rapid Acting Intra-Muscular Olanzapine in Japanese Patients With Schizophrenia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5293; F1D-JE-RA01
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — olanzapine-fluoxetine combination

INTERVENTIONS:
Drug: Olanzapine Hydrochloride

SUMMARY:
The purpose of this study is to examine the clinical therapeutic dose in Japanese agitated patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 20 years of age and less than 65 years old
* Patients must be inpatients during the study
* Patients must have a diagnosis of schizophrenia as per the DSM-IV, as determined by the investigator
* Patients must be considered by the investigator to be clinically agitated and to be clinically appropriate candidates for the treatment with intramuscular (IM) medication
* Patients must have a minimum total score of greater than or equal to 14 on the 5 items of the PANSS-EC and at least one individual item score of greater than or equal to 4 using the 1-7 scoring system, prior to the first IM injection of study drug

Exclusion Criteria:

* Serious, unstable illnesses such that death is anticipated within 1 year or intensive care unit hospitalization for the disease is anticipated within 6 months. This includes hepatic (specifically any degree of jaundice), renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic diseases
* Known history of seizures; however, a patient whose etiology is identifiable and has been resolved may be enrolled
* Known history of diabetes mellitus, complications of diabetes mellitus, or potential diabetes mellitus as defined by patients with single blood glucose measurement based on site tests; patients with values greater than or equal to 140 mg/dL (non-fasting) or greater than or equal to 110 mg/dL (fasting) must be excluded from the study
* History of allergic reaction or intolerance to olanzapine
* Have received treatment with psychostimulants or reserpine within 1 week prior to study drug administration

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2004-06; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
The primary objective is to examine the safety and efficacy of the clinical therapeutic dose of IM olanzapine (7.5 mg/inj and 10 mg/inj) in Japanese agitated patients with schizophrenia

SECONDARY OUTCOMES:
To examine the efficacy of IM olanzapine by evaluating change from baseline to 24 hours following the first IM injection in the PANSS Excited Component Total Score and the ACES
To examine the characteristics of sedation for each treatment group based on the ACES score
To examine a frequency of patients who needed second injection

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo, Japan

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com